CLINICAL TRIAL: NCT01020539
Title: Allogeneic Stem Cell Transplantation Followed By Targeted Immune Therapy In Average Risk Acute Myelogenous Leukemia/Myelodysplastic Syndrome/Juvenile Myelomonocytic Leukemia (AML/MDS/JMML)
Brief Title: Allogeneic Stem Cell Transplantation Followed By Targeted Immune Therapy In Average Risk Leukemia
Acronym: AML/MDS/JMML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Monica Bhatia, Associate Professor of Pediatrics, Section Head of Pediatric Stem Cell Transplant at Columbia University, Columbia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA6378; CHNY-504 (Other: CU)
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Juvenile Myelomonocytic Leukemia
Keywords: Allogeneic Stem Cell Transplantation; Targeted Immune Therapy; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Juvenile Myelomonocytic Leukemia; AML; MDS; JMML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Juvenile | interventions — fludarabine; fludarabine phosphate; Busulfan; Gemtuzumab; Antilymphocyte Serum; thymoglobulin; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Matched Family Donor (Experimental): Patients will receive a reduced intensity fludarabine (6 days)/busulfan (2 days) conditioning regimen followed by a stem cell transplant from a related family donor using bone marrow or cord blood stem cells. Then followed by Gemtuzumab Ozogamicin, once at about 2-6 months post alloSCT and once at least 2 months after the first dose. Patients with JMML will also receive cis-retinoic acid (Isotretinoin).
  During and following transplantation patients will receive methylprednisolone for immune suppression. Graft-versus-host-disease (GVHD) prophylaxis will consist of tacrolimus, mycophenolate mofetil and additionally methotrexate in recipients of unrelated adult transplants.
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: GVHD Prophylaxis; Drug: Gemtuzumab Ozogamicin
- Unrelated Donor (Experimental): Patients will receive a reduced intensity fludarabine (6 days)/busulfan (2 days) conditioning regimen followed by a stem cell transplant from an unrelated donor using matched bone marrow or cord blood stem cells.Then followed by Gemtuzumab Ozogamicin, once at about 2-6 months post alloSCT and once at least 2 months after the first dose. Patients with JMML will also receive cis-retinoic acid (Isotretinoin).
  During and following transplantation patients will receive methylprednisolone for immune suppression and unrelated donor transplant recipients will additionally receive Anti-Thymocyte Globulin. GVHD prophylaxis will consist of tacrolimus, mycophenolate mofetil and additionally methotrexate in recipients of unrelated adult transplants.
  Interventions: Drug: Anti-Thymocyte Globulin; Drug: Isotretinoin

INTERVENTIONS:
Drug: Fludarabine — Conditioning Regimen
  Other Names: Fludara®
  Arms: Matched Family Donor
Drug: Busulfan — Conditioning Regimen
  Other Names: Busulfex®
  Arms: Matched Family Donor
Drug: GVHD Prophylaxis — Can be FK506 (Tacrolimus/Prograf®), mycophenolate mofetil ((MMF)/Cellcept®), or methotrexate (MTX, amethopterin)
  Arms: Matched Family Donor
Drug: Gemtuzumab Ozogamicin — Dose Escalation
  Other Names: Mylotarg®
  Arms: Matched Family Donor
Drug: Anti-Thymocyte Globulin — Unrelated Donors only
  Other Names: Thymoglobulin®
  Arms: Unrelated Donor
Drug: Isotretinoin — JMML patients only
  Other Names: Accutane®; 13-cis-Retinoic Acid (cis-RA)
  Arms: Unrelated Donor

SUMMARY:
Allogeneic stem cell transplantation (AlloSCT) followed by targeted immune therapy Gemtuzumab Ozogamicin patients with acute myeloid leukemia (AML)/juvenile myelomonocytic leukemia (JMML)/myelodysplastic syndromes (MDS) will be safe and well tolerated.

DETAILED DESCRIPTION:
Gemtuzumab Ozogamicin (CMA-676) is a chemotherapeutic agent consisting of a recombinant humanized anti-CD33 antibody conjugated with calicheamicin, a highly potent cytotoxic antitumor antibiotic. The antibody portion of Gemtuzumab binds specifically to the CD33 antigen, a sialic acid-dependent adhesion protein expressed on the surface of leukemic blasts, normal and leukemic myeloid colony-forming cells, including leukemic clonogenic precursors, but excluding pluripotent hematopoietic stem cells and nonhematopoietic cells. This results in formation of a complex that is internalized, upon which the calicheamicin derivative is released within the lysosomes of the myeloid cell. The free calicheamicin derivative then binds to deoxyribonucleic acid (DNA), resulting in DNA double strand breaks and consequential cell death. Over 80% of AML patients possess myeloid blast cells with CD33 surface antigen expression.

ELIGIBILITY:
Inclusion Criteria:

Disease Status

* AML 1st complete remission (CR) with a matched family donor (excluding Downs Syndrome, acute promyelocytic leukaemia (APL), poor cytogenetics (12p, 5q, -7 and FMS-like tyrosine kinase 3 (FLT3) mutations or duplication t(9;11) and others)) and patients consented to and registered on an upfront AML COG study with a matched family donor)
* AML 1st CR (excluding Downs Syndrome, APL, and chromosome translocation (8;21) or inversion (16) or poor cytogenetics (12p, 5q, -7, FLT3 mutation or duplication t(9;11) and others)) with unrelated donor
* AML 2nd CR
* Myelodysplastic Syndrome (MDS) and ≤ 5% bone marrow myeloblasts at diagnosis (de novo patients only)
* Juvenile Myelomonocytic Leukemia (JMML) and ≤ 5% bone marrow myeloblasts at diagnosis

In regards to disease immunophenotype, disease must express a minimum of ≥10% Cell Differential 33 (CD33) positivity for patients with AML

Organ Function:

Patients must have adequate organ function as defined below:

Adequate renal function defined as:

* Serum creatinine < 1.5 x normal, or
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) 40 ml/min/m2 or > 60 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range

Adequate liver function defined as total bilirubin 2.0 x upper limit of normal (ULN), or serum glutamic-oxaloacetic transaminase (SGOT)(aspartate aminotransferase (AST)) or serum glutamic-pyruvic transaminase (SGPT)(alanine aminotransferase (ALT)) < 5.0 x ULN

Adequate cardiac function defined as:

* Shortening fraction of ≥ 25% by echocardiogram, or
* Ejection fraction of ≥ 45% by radionuclide angiogram or echocardiogram

Adequate pulmonary function defined as:

* Diffusion capacity of the lung for carbon monoxide (DLCO) ≥ 40% by pulmonary function tests (PFT) (Uncorrected)
* For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% on room air

Exclusion Criteria:

* Patients with active central nervous system (CNS) AML/JMML disease at time of preparative regimen
* Secondary MDS
* Poor cytogenetics (12p, 5q, -7, FLT3 mutation or duplication)
* Female patients who are pregnant (positive human chorionic gonadotropin(hCG))
* Karnofsky <70% or Lansky <50% if 10 years or less
* Age >30 years
* Seropositive for Human Immunodeficiency Virus (HIV)
* Patients consented to and registered on an upfront Children's Oncology Group (COG) AML study with a matched family donor

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2002-09-11 (Actual); Primary Completion 2011-07-20 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated and/or biologically active dose of Gemtuzumab Ozogamicin (GO) | Up to 2 years
  To determine the maximal tolerated and/or biologically active dose of Gemtuzumab Ozogamicin (GO) (anti CD33 immunotoxin) therapy following reduced intensity (RI) allogeneic stem cell transplantation (alloSCT) in patients with average risk AML/JMML/MDS.

SECONDARY OUTCOMES:
Change of minimal residual disease | Day 60, Day 100, Day 180, 1 year, 2 years
  To measure the changes, if applicable, of minimal residual disease prior to and after consolidation therapy with targeted immunotherapy in average risk AML/JMML/MDS post RI AlloSCT.
Incidence of minor histocompatibility antigen (MHA) expression on acute myeloid leukemia (AML) tissue | Up to 2 years
  To measure the minor histocompatibility antigen expression on AML tissue, donor and recipient, and the incidence of development of MHA specific cytotoxic T-lymphocytes (CTLs).
Degree of mixed/complete donor chimerism | Up to 2 years
  To determine the degree of mixed/complete donor chimerism after RI AlloSCT in patients with average risk AML/JMML/MDS.
Event free survival (EFS) rate | Up to 2 years
  To determine event free survival (EFS) after RI AlloSCT and targeted immunotherapy in patients with average risk AML/JMML/MDS.
Overall survival (OS) rate | Up to 2 years
  To determine overall survival (OS) after RI AlloSCT and targeted immunotherapy in patients with average risk AML/JMML/MDS.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bhatia, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided